CLINICAL TRIAL: NCT06988774
Title: Assessment of Tubal Occlusion During Minimally Invasive Myomectomy
Acronym: ATOM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00008836
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Fallopian Tube Patency Tests; Fibroid/Myoma (Uterus/Cervix); Myomectomy; Fallopian Tube Disease
Keywords: chromopertubation; myomectomy; uterine fibroids; fallopian tube disease
MeSH Terms: conditions — Leiomyoma; Myoma; Fallopian Tube Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ATOM study participants (Experimental): Patients enrolled in the study who will undergo the chromopertubation per protocol
  Interventions: Procedure: chromopertubation

INTERVENTIONS:
Procedure: chromopertubation — Pre- and post-myomectomy chromopertubation procedure using dilute methylene blue dye solution for evaluation of tubal occlusion

SUMMARY:
This study uses a procedure called chromopertubation to look at how fibroids and fibroid surgery affect the fallopian tubes. Specifically, this study will test if the fallopian tubes are occluded or patent (open) before and after surgically removing fibroids.

Chromopertubation is a commonly performed and well-established procedure that is done during laparoscopic surgery to determine if the fallopian tubes are open or blocked. It includes inserting a dilute solution of saline with a small amount of medical-grade blue dye (called methylene blue) into the uterine cavity to see if it spills out of the fallopian tubes. Chromopertubation is considered a safe procedure - the main risk is an allergic reaction to the dye, which is very rare. The minimum amount of methylene blue dye will be used to further reduce risks of a reaction.

Open fallopian tubes are necessary to become pregnant without the use of IVF. While it is known that some conditions can affect the functioning of the fallopian tubes, there is a lack of research about how fibroids affect the tubes. It is also not known how much about how the process of removing fibroids may affect the fallopian tubes. The investigators hypothesize that tubal occlusion will be observed in patients with fibroids and that the frequency of tubal occlusion will change after myomectomy compared to pre-myomectomy.

This study will be conducted entirely during planned surgery for laparoscopic myomectomy. Chromopertubation will be performed at the beginning and again at the end of the surgery. This is expected to take less than 10 minutes in total. The results of the chromopertubation as well as background medical information will be recorded and the characteristics of the fibroids (size, number, and location) will be compared to the presence or abscence of tubal occlusion as determined by chromopertubation.

DETAILED DESCRIPTION:
Background:

Fibroids have a prevalence >75%, making it the most common benign uterine disease [Zepiridis 2016, Lazaridis 2013, Giuliani 2020]. Fibroids are well known to contribute to infertility and early pregnancy loss [Don 2023, Pritts 2025, Carson 2021, Giuliani 2020]. This is typically thought to be secondary to distortion and impairment of the endometrial cavity or myometrial junction. However, it has been stressed in recent reviews that the full mechanism of the effect of fibroids on infertility is not fully understood, and more studies are needed [Donnez 2024]. It is theorized but not well confirmed through evidence-based studies that fibroids may also occlude or compress fallopian tubes and contribute to tubal occlusion that may contribute to infertility [Don 2023, Zepiridis 2016, Horne 2007, Somigliana 2021]. Additionally, up to 25-35% of female-factor infertility is related to tubal disease [ASRM Practice Committee 2021, Carson 2021, Mayrhofer 2022]. There is very little data on tubal patency assessment in patients undergoing myomectomy. The investigators have been able to identify only one prospective study from 1993 that specifically evaluated fallopian tube filling during post-myomectomy hysterosalpingogram, though the primary outcome of this study was endometrial cavity architecture [Lev-Toaff 1993]. Two recent retrospective studies have demonstrated a significant association between presence of leiomyoma and tubal occlusion in women with infertility [Mayrhofr 2024, Nako 2024]. Nako et al (2024) found a significant association only with submucosal fibroids. The investigators have not identified any recent prospective studies evaluating tubal patency in patients with uterine leiomyoma or those undergoing myomectomy.

Most data regarding tubal patency assessment are collected on patients already diagnosed with infertility, which introduces the possibility of multiple confounding variables. There are no recent prospective studies of tubal occlusion in patients with fibroids or patients undergoing myomectomy.

Earlier detection of tubal disease may allow for a quicker and more proactive work up and counseling before other factors such as age and oocyte quality further impact fertility options. There is also limited data on tubal occlusion or patency in patients with fibroids and those undergoing myomectomy. Underappreciation of the effect of uterine fibroids and myomectomy on tubal patency and subsequent delays in diagnosis could further complicate fertility due to age, reduced ovarian reserve and oocyte quality. Knowledge of tubal occlusion may influence referral to an infertility specialist or counseling for ectopic pregnancy risk.

Objectives:

To evaluate the incidence of tubal occlusion in patients undergoing surgery for uterine fibroids before and after surgical intervention.

To assess the correlation between tubal patency and fibroid characteristics based on FIGO classification in patients undergoing surgery for uterine fibroids.

To assess characteristics of patients who have change in tubal occlusion.

This proposed study can help contribute to a more proactive approach to early detection and intervention for tubal occlusion in a high-risk patient population in order to achieve the following goals: to improve understanding of the effects of fibroids and myomectomy on tubal occlusion and to gain a better understanding in order to inform future studies to optimize counseling, diagnosis, and early intervention for tubal occlusive disease.

Design:

This is a single-arm prospective study using chromopertubation to assess tubal occlusion in patients undergoing minimally invasive gynecologic surgery for uterine fibroids. This procedure involves injecting a dilute solution of medical-grade dye into the endometrial cavity and visualizing spillage of the dye through the fallopian tubes into the abdominal cavity, indicating patency of the tubes that would allow for spontaneous conception. Chromopertubation will be performed at the initiation and completion of the surgery and tubal occlusion will be documented.

Chromopertubation procedure:

Pre-surgery: chromopertubation will be performed at the start of laparoscopic or robotic surgical procedure, once abdominal ports are in place and uterine manipulator placement has been performed prior to initiation of any myomectomy or other interventional surgical procedures.

Post-surgery: Chromopertubation will again be performed at the end of the surgery, once all surgical interventions are complete and prior to removal of abdominal ports and uterine manipulator.

Chromopertubation will be performed per standard clinical protocol as follows: Up to 50 mL of dilute methylene blue dye solution (1mL of 10 mg/mL 1% methylene blue in 200 mL normal saline) will be injected into the uterine cavity through a uterine manipulator with a patent central channel. This dose totals up to 2.5 mg of dilute methylene blue dye per chromopertubation injection and an anticipated maximum dose of 5 mg of dilute methylene blue per patient. Spillage of dye should be visible immediately after injection of dilute dye into the endometrial cavity if tubes are patent.

Adverse event monitoring:

As chromopertubation is an established medical procedure, patients will be monitored according to the standard intra-operative and post-operative criteria. If there are any signs of adverse events prior to completion of the study interventions, the study procedure will be aborted immediately and supportive therapy provided as needed. This will be done through communication between the surgical and anesthesiology teams.

Patients will be observed in the post-anesthesia care unit (PACU) according to standard postoperative protocol for any adverse events. In accordance with our standard post-operative practice, all patients will be discharged home upon meeting standard postoperative discharge criteria. As per routine standard protocol, all patients will be called at home to assess for any issues or concerns and to see how they are doing overall. This call is performed by either the attending surgeon or fellow on post-operative day #1, if discharged after surgery, or rounded on if admitted to the hospital overnight. Patients who report adverse effects once at home will be triaged and evaluated according to standard post-operative precautions.

There are no plans for long-term follow up at this time. Data will be collected intraoperatively and from chart review, including

* Pre-myomectomy tubal patency or occlusion - unilateral vs bilateral, proximal vs distal
* Post-myomectomy tubal patency or occlusion - unilateral vs bilateral, proximal vs distal
* Size, anatomic location and FIGO classification of fibroids removed
* Number of fibroids removed and total weight in grams
* Presence of endometriosis diagnosed intraoperatively
* Patient age, medical, surgical, obstetric, and gynecologic history
* Pre-operative imaging reports of the uterus/fibroids

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing minimally invasive laparoscopic or robotic-assisted uterine-preserving gynecologic surgery for removal of uterine fibroids (myomectomy) by a minimally invasive gynecologic surgeon at MedStar.

Exclusion Criteria:

* Patients with both fallopian tubes absent
* Patients in whom it is not possible to place a uterine manipulator or catheter
* Patient with known tubal disease or occlusion, or patients who have undergone prior tubal surgery
* Patients with allergy to methylene blue dye or G6PD deficiency
* Patients with positive pregnancy test on day of surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of tubal occlusion pre- and post-myomectomy | Limited to the duration of each surgery
  Frequency of tubal occlusion in patients with fibroids immediately prior to and after completion of myomectomy procedures. Spillage of methylene blue dye seen laparoscopically is indicative of tubal patency. Unilateral vs bilateral occlusion will be documented.

SECONDARY OUTCOMES:
Frequency of tubal occlusion compared to fibroid characteristics | Limited to the duration of each surgery
  Frequency of tubal occlusion as compared to fibroid(s):
  * FIGO classification
  * size
  * anatomic location
Change in tubal occlusion | Limited to the duration of each surgery
  Frequency of change in tubal occlusion comparing pre-myomectomy to post-myomectomy. Ex. occluded to patent or patent to occluded.

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbieri RL. Farewell to indigo carmine. OBG Management. 2014. https://mdedge.com/obgmanagement/article/86698/pelvic-floor-dysfunction/farewell-indigo-carmine.
- [Background] Zepiridis LI, Grimbizis GF, Tarlatzis BC. Infertility and uterine fibroids. Best Pract Res Clin Obstet Gynaecol. 2016 Jul;34:66-73. doi: 10.1016/j.bpobgyn.2015.12.001. Epub 2015 Dec 23. PMID 26856931
- [Background] Somigliana E, Reschini M, Bonanni V, Busnelli A, Li Piani L, Vercellini P. Fibroids and natural fertility: a systematic review and meta-analysis. Reprod Biomed Online. 2021 Jul;43(1):100-110. doi: 10.1016/j.rbmo.2021.03.013. Epub 2021 Mar 23. PMID 33903032
- [Background] Saunders RD, Shwayder JM, Nakajima ST. Current methods of tubal patency assessment. Fertil Steril. 2011 Jun;95(7):2171-9. doi: 10.1016/j.fertnstert.2011.02.054. Epub 2011 Mar 31. PMID 21457959
- [Background] Sankey-Thomas KM, Travieso J, Salazar CA, Williams-Brown M, Breen MT. Fertility sparing management of a large broad ligament fibroid. Journal of Minimally Invasive Gynecology. 2024;31(11, Supplement):S6.
- [Background] Rzymski P, Wozniak J, Opala T, Wilczak M, Sajdak S. Anaphylactic reaction to methylene blue dye after laparoscopic chromopertubation. Int J Gynaecol Obstet. 2003 Apr;81(1):71-2. doi: 10.1016/s0020-7292(03)00036-5. No abstract available. PMID 12676403
- [Background] Ramin S, Azar FP, Malihe H. Methylene blue as the safest blue dye for sentinel node mapping: emphasis on anaphylaxis reaction. Acta Oncol. 2011 Jun;50(5):729-31. doi: 10.3109/0284186X.2011.562918. Epub 2011 Mar 17. No abstract available. PMID 21413854
- [Background] Pritts EA, Parker WH, Olive DL. Fibroids and infertility: an updated systematic review of the evidence. Fertil Steril. 2009 Apr;91(4):1215-23. doi: 10.1016/j.fertnstert.2008.01.051. Epub 2008 Mar 12. PMID 18339376
- [Background] Nako Y, Ota K, Sujino T, Mitsui J, Kamo H, Katsumata S, Takayanagi Y, Tajima M, Ishikawa T, Komiya A, Kawai K. A Large Study About Reproductive Factors That Predict Hysterosalpingography-Identified Tubal Pathology: An Insight into the Necessity of Preconception Screening. J Clin Med. 2024 Dec 31;14(1):179. doi: 10.3390/jcm14010179. PMID 39797266
- [Background] Mayrhofer D, Parry JP, Hager M, Beitl K, Kurz C, Ott J. Are the Stage and the Incidental Finding of Endometriosis Associated with Fallopian Tube Occlusion? A Retrospective Cohort Study on Laparoscopic Chromopertubation in Infertile Women. J Clin Med. 2022 Jun 28;11(13):3750. doi: 10.3390/jcm11133750. PMID 35807038
- [Background] Mayrhofer D, Holzer I, Aschauer J, Selzer C, Parry JP, Ott J. Incidence and Causes of Tubal Occlusion in Infertility: A Retrospective Cohort Study. J Clin Med. 2024 Jul 6;13(13):3961. doi: 10.3390/jcm13133961. PMID 38999525
- [Background] Lev-Toaff AS, Karasick S, Toaff ME. Hysterosalpingography before and after myomectomy: clinical value and imaging findings. AJR Am J Roentgenol. 1993 Apr;160(4):803-7. doi: 10.2214/ajr.160.4.8456668.
- [Background] Lazaridis A, Hirsch M, Pistofidis G, Odejinmi F. Surgical management of uterine fibroids. Curr Opin Obstet Gynecol. 2023 Oct 1;35(5):440-445. doi: 10.1097/GCO.0000000000000903. Epub 2023 Aug 2. PMID 37548229
- [Background] Jena SK, Naik SS. Methemoglobinaemia after diagnostic hystero-laparoscopic chromopertubation in a sub-fertile patient. J Obstet Gynaecol. 2019 Oct;39(7):1025-1026. doi: 10.1080/01443615.2019.1581744. Epub 2019 Jun 9. No abstract available. PMID 31179795
- [Background] Horne AW, Critchley HO. The effect of uterine fibroids on embryo implantation. Semin Reprod Med. 2007 Nov;25(6):483-9. doi: 10.1055/s-2007-991046. PMID 17960533
- [Background] Giuliani E, As-Sanie S, Marsh EE. Epidemiology and management of uterine fibroids. Int J Gynaecol Obstet. 2020 Apr;149(1):3-9. doi: 10.1002/ijgo.13102. Epub 2020 Feb 17. PMID 31960950
- [Background] Egbe TO, Nana-Njamen T, Elong F, Tchounzou R, Simo AG, Nzeuga GP, Njamen Nana C, Manka'a E, Tchente Nguefack C, Halle-Ekane GE. Risk factors of tubal infertility in a tertiary hospital in a low-resource setting: a case-control study. Fertil Res Pract. 2020 Mar 6;6:3. doi: 10.1186/s40738-020-00073-4. eCollection 2020. PMID 32161654
- [Background] Donnez J, Taylor HS, Marcellin L, Dolmans MM. Uterine fibroid-related infertility: mechanisms and management. Fertil Steril. 2024 Jul;122(1):31-39. doi: 10.1016/j.fertnstert.2024.02.049. Epub 2024 Mar 5. PMID 38453041
- [Background] Don EE, Mijatovic V, Huirne JAF. Infertility in patients with uterine fibroids: a debate about the hypothetical mechanisms. Hum Reprod. 2023 Nov 2;38(11):2045-2054. doi: 10.1093/humrep/dead194. PMID 37771247
- [Background] Carson SA, Kallen AN. Diagnosis and Management of Infertility: A Review. JAMA. 2021 Jul 6;326(1):65-76. doi: 10.1001/jama.2021.4788. PMID 34228062
- [Background] Bezu C, Coutant C, Salengro A, Darai E, Rouzier R, Uzan S. Anaphylactic response to blue dye during sentinel lymph node biopsy. Surg Oncol. 2011 Mar;20(1):e55-9. doi: 10.1016/j.suronc.2010.10.002. Epub 2010 Nov 11. PMID 21074413
- [Background] Bagadia R, Kanabar V. Can laparoscopic chromopertubation with methylene blue dye cause anaphylactic reactions like pulmonary edema? WJOLS. 2017;10(2):51-53.
- [Background] Practice Committee of the American Society for Reproductive Medicine. Electronic address: ASRM@asrm.org. Role of tubal surgery in the era of assisted reproductive technology: a committee opinion. Fertil Steril. 2021 May;115(5):1143-1150. doi: 10.1016/j.fertnstert.2021.01.051. Epub 2021 Feb 26. PMID 33642065
- [Background] Ansari AH. Methylene blue test for assessment of tubal patency: a new and simple technique. Can Med Assoc J. 1968 Jul 27;99(4):182-4. No abstract available. PMID 5317820
- [Background] Akazawa M, Wu YH, Liu WM. Allergy-like reactions to methylene blue following laparoscopic chromopertubation: A systematic review of the literature. Eur J Obstet Gynecol Reprod Biol. 2019 Jul;238:58-62. doi: 10.1016/j.ejogrb.2019.03.019. Epub 2019 Mar 20. PMID 31112852

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT06988774/Prot_SAP_000.pdf
  • Informed Consent Form (2025-05-16): https://cdn.clinicaltrials.gov/large-docs/74/NCT06988774/ICF_001.pdf